CLINICAL TRIAL: NCT05954650
Title: Minimally Conscious State Plus Versus Minus: Likelihood of Emergence and Long-term Functional Independence
Brief Title: Clinical Validity of the Minimally Conscious State "Plus" and "Minus"
Status: Completed | Type: Observational
Sponsor: Hospitales Nisa (Other)
Collaborators: Generalitat Valenciana (Other)
Responsible Party: Sponsor
Other Study IDs: P0428112022
Record Dates: First submitted 2023-07-06; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Disorder of Consciousness
Keywords: Disorders of Consciousness; Minimally Conscious State; Minimally Conscious State Plus; Minimally Conscious State Minus; Disability Rating Scale; Functional Independence
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in a Minimally Conscious State: Patients diagnosed as in a Minimally Conscious State "Plus" and "Minus"
  Interventions: Behavioral: Rehabilitation

INTERVENTIONS:
Behavioral: Rehabilitation — Physical therapy and multisensory stimulation adjusted to the needs of each patient.

SUMMARY:
The goal of this observational retrospective study is to investigate and compare the clinical evolution of a sample of patients with the diagnosis of MCS+ versus MCS- according to the CRS-R. The main questions it aims to answer are the presence of differences in the likelihood of emergence from the MCS (EMCS) between these two groups and in the progress of disability and functional independence after the EMCS.

DETAILED DESCRIPTION:
Severe acquired brain injuries can be caused by traumatic brain injury, stroke or anoxia, among others and can lead to Disorders of Consciousness (DOC), an umbrella term that encompasses a wide range of different clinical conditions such as coma, the Unresponsive Wakefulness Syndrome (UWS) and the Minimally Conscious State (MCS). Coma usually lasts from a few days to few weeks and it is defined as a state of profound unawareness from which the patient cannot be aroused; eyes are closed, and a normal sleep-wake cycle is absent. The UWS denotes a condition of wakefulness without (clinical signs of) awareness; UWS patients may open their eyes but exhibit only reflex (i.e. non-intentional) behaviors and are therefore considered unaware of themselves and their surroundings. On the other hand, the MCS denotes a condition where discernible behavioral evidence of consciousness is retained. More recently, given the heterogeneity of the MCS category, patients showing higher level responses, including reproducible movements to commands, intelligible verbalization and intentional communication (i.e. MCS+), have been distinguished from those showing lower level non-reflex responses (e.g. visual pursuit, object recognition; i.e. MCS-). Once patients recovery the ability to communicate or to use objects they are considered emerged from the MCS (EMCS).

Currently, the gold standard for the behavioural assessment of DOC patients is the Coma Recovery Scale-Revised (CRS-R) and the diagnosis is made according to the presence of certain behaviours. However, because of daily fluctuations, a minimum of 5 CRS-R evaluations within a short time interval are recommended, allowing to reduce the risk of misdiagnose to the 40%.

If the CRS-R criteria for the diagnosis of coma and UWS are somehow clear, the MCS and EMCS entities are the focus of a growing body of research. Despite all, the diagnostic criteria for DOC patients are becoming clearer and clearer, but markers to predict prognosis and functional outcome need to be better studied. Knowing the natural history of patients with DOC may help to an adequate prognosis, that is important not only for the patient and the family but also for treatment planning and provision of therapies and discharge. In particular, if there are existing studies about the prognosis of UWS and MCS patients, studies comparing MCS- and MCS+ patients are lacking. State of the art about the prognosis in DOC patients highlight a better outcome for patients in a MCS compared to patients in UWS, but little is known about a possible different prognosis between MCS+ and MCS- patients. A recent study stresses the need for prospective studies investigating differences in long-term functional outcome between patients in a MCS+ and MCS-. So far, the only available longitudinal study including MCS- and MCS+ patients followed 39 chronic DOC patient for two years after brain injury and assessed them with the CRS-R every 3 months. The sample included 16 patients in a UWS, 15 patients in a MCS-, 7 in a MCS+ and 1 in a EMCS and the authors did not find differences in the prognosis between MCS- and MCS+ patients, probably due to limited sample size.

Therefore, the first aim of this study is to investigate and compare the clinical evolution of a sample of patients with the diagnosis of MCS+ versus MCS- according to the CRS-R total score. In particular, the investigators focus our attention on the likelihood of emergence from the MCS and on the evolution of functional independence after the emergence from the MCS. The investigators hypothesize that those patients presenting preferentially complex behavioural responses will have better clinical trajectories including an increasing likelihood to emerge form MCS and a better functional outcome once emerged from the MCS.

ELIGIBILITY:
Inclusion Criteria:

* Severe acquired brain injury leading to a Disorder of Consciousness (DOC)
* Persistance of the DOC for a period not inferior to 28 days and not longer than 6 months
* Diagnosis of MCS
* Having a fa follow-up period of no less than 12 months from the onset

Exclusion Criteria:

* Diagnosis of UWS
* Being younger than 18 years
* DOC persisting more than 6 months
* Absence of follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data of patients with DOC who had attended an inpatient neurorehabilitation program between January 2004 and December 2022 in all facilities of the hospital network.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2004-09-30 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Baseline clinical state | At admission to the rehabilitation hospital
  Defined by the clinical state (Unresposive Wakefulness Syndrome, Minimally Conscious State, Emergence from Minimally Conscious State).
Baseline neurobehavioral condition | At admission to the rehabilitation hospital
  Defined by the score in the Coma Recovery Scale-Revised (CRS-R).
  The CRS-R consists of 29 hierarchically organised items divided into 6 subscales addressing auditory, visual, motor, oromotor, communication, and arousal processes.
Baseline disability | At the admission to the rehabilitation hospital
  Defined by scores in the Disability Rating Scale (DRS).
  The DRS is an 8-item scale that address the three original World Health Organization categories of impairment, disability and handicap. Scores obtained from the Disability Rating Scale can be interpreted as indicators of various levels of disability, including no disability (score of 0), mild (1), partial (2-3), moderate (4-6), moderately severe (7-11), severe (12-16), extremely severe (17-21), vegetative state (22-24), and extreme vegetative state (25-29).
Progress in the clinical state | Weekly assessments from admission to the rehabilitation hospital to discharge, demise, or emergence from MCS, up to 36 months
  Defined by the clinical state (Unresposive Wakefulness Syndrome, Minimally Conscious State, Emergence from Minimally Conscious State).
Progress in the neurobehavioral condition | Weekly assessments from admission to the rehabilitation hospital to discharge, demise, or emergence from MCS, up to 36 months
  Defined by the score in the Coma Recovery Scale-Revised (CRS-R).
  The CRS-R consists of 29 hierarchically organised items divided into 6 subscales addressing auditory, visual, motor, oromotor, communication, and arousal processes.
Progress in disability | Monthly assessments from admission to the rehabilitation hospital to discharge, demise, or emergence from MCS, up to 36 months
  Defined by scores in the Disability Rating Scale (DRS).
  The DRS is an 8-item scale that address the three original World Health Organization categories of impairment, disability and handicap. Scores obtained from the Disability Rating Scale can be interpreted as indicators of various levels of disability, including no disability (score of 0), mild (1), partial (2-3), moderate (4-6), moderately severe (7-11), severe (12-16), extremely severe (17-21), vegetative state (22-24), and extreme vegetative state (25-29).
Follow-up disability | At 6 months after emergence from MCS
  Defined by scores in the Disability Rating Scale (DRS).
  The DRS is an 8-item scale that address the three original World Health Organization categories of impairment, disability and handicap. Scores obtained from the Disability Rating Scale can be interpreted as indicators of various levels of disability, including no disability (score of 0), mild (1), partial (2-3), moderate (4-6), moderately severe (7-11), severe (12-16), extremely severe (17-21), vegetative state (22-24), and extreme vegetative state (25-29).
Follow-up independence in activities of daily living | At 6 months after emergence from MCS
  Defined by scores in the Barthel Index (BI).
  The BI measures the degree of assistance required by an individual on 10 items of mobility and self care. The scores in the BI can be interpreted as indicators of dependence, such as total dependence (scores below 21), severe dependence (21-60), moderate dependence (61-90), and slight dependence (scores above 90).
Follow-up functional Independence | At 6 months after emergence from MCS
  Defined by scores in the Functional Independence Measure (FIM).
  The FIM is a 18-item that measures independence for self-care, including sphincter control, transfers, locomotion, communication, and social cognition. The total score of the FIM can be interpreted as a general measure of functional independence and also as stages of functional independence within activities of daily living, sphincter management, mobility, and executive function.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospitales NISA, Valencia
  - Servicio de Neurorrehabilitación y Daño Cerebral de los Hospitales NISA, Valencia

REFERENCES:
- [Background] Bareham CA, Allanson J, Roberts N, Hutchinson PJA, Pickard JD, Menon DK, Chennu S. Longitudinal assessments highlight long-term behavioural recovery in disorders of consciousness. Brain Commun. 2019;1(1):fcz017. doi: 10.1093/braincomms/fcz017. Epub 2019 Sep 16. PMID 31886461
- [Background] Bruno MA, Vanhaudenhuyse A, Thibaut A, Moonen G, Laureys S. From unresponsive wakefulness to minimally conscious PLUS and functional locked-in syndromes: recent advances in our understanding of disorders of consciousness. J Neurol. 2011 Jul;258(7):1373-84. doi: 10.1007/s00415-011-6114-x. Epub 2011 Jun 16. PMID 21674197
- [Background] Bruno MA, Majerus S, Boly M, Vanhaudenhuyse A, Schnakers C, Gosseries O, Boveroux P, Kirsch M, Demertzi A, Bernard C, Hustinx R, Moonen G, Laureys S. Functional neuroanatomy underlying the clinical subcategorization of minimally conscious state patients. J Neurol. 2012 Jun;259(6):1087-98. doi: 10.1007/s00415-011-6303-7. Epub 2011 Nov 12. PMID 22081100
- [Background] Colantonio A, Gerber G, Bayley M, Deber R, Yin J, Kim H. Differential profiles for patients with traumatic and non-traumatic brain injury. J Rehabil Med. 2011 Mar;43(4):311-5. doi: 10.2340/16501977-0783. PMID 21347507
- [Background] Katz DI, Polyak M, Coughlan D, Nichols M, Roche A. Natural history of recovery from brain injury after prolonged disorders of consciousness: outcome of patients admitted to inpatient rehabilitation with 1-4 year follow-up. Prog Brain Res. 2009;177:73-88. doi: 10.1016/S0079-6123(09)17707-5. PMID 19818896
- [Background] Giacino JT, Ashwal S, Childs N, Cranford R, Jennett B, Katz DI, Kelly JP, Rosenberg JH, Whyte J, Zafonte RD, Zasler ND. The minimally conscious state: definition and diagnostic criteria. Neurology. 2002 Feb 12;58(3):349-53. doi: 10.1212/wnl.58.3.349. PMID 11839831
- [Background] Giacino JT, Kalmar K, Whyte J. The JFK Coma Recovery Scale-Revised: measurement characteristics and diagnostic utility. Arch Phys Med Rehabil. 2004 Dec;85(12):2020-9. doi: 10.1016/j.apmr.2004.02.033. PMID 15605342
- [Background] Golden K, Erler KS, Wong J, Giacino JT, Bodien YG. Should Consistent Command-Following Be Added to the Criteria for Emergence From the Minimally Conscious State? Arch Phys Med Rehabil. 2022 Sep;103(9):1870-1873. doi: 10.1016/j.apmr.2022.03.010. Epub 2022 Apr 6. PMID 35398046
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Pape TL, Lundgren S, Heinemann AW, Guernon A, Giobbie-Hurder A, Wang J, Roth H, Blahnik M, Williams V. Establishing a prognosis for functional outcome during coma recovery. Brain Inj. 2006 Jun;20(7):743-58. doi: 10.1080/02699050600676933. PMID 16809207
- [Background] Rappaport M, Hall KM, Hopkins K, Belleza T, Cope DN. Disability rating scale for severe head trauma: coma to community. Arch Phys Med Rehabil. 1982 Mar;63(3):118-23. PMID 7073452
- [Background] Song M, Yang Y, Yang Z, Cui Y, Yu S, He J, Jiang T. Prognostic models for prolonged disorders of consciousness: an integrative review. Cell Mol Life Sci. 2020 Oct;77(20):3945-3961. doi: 10.1007/s00018-020-03512-z. Epub 2020 Apr 18. PMID 32306061
- [Background] Stineman MG, Ross RN, Fiedler R, Granger CV, Maislin G. Functional independence staging: conceptual foundation, face validity, and empirical derivation. Arch Phys Med Rehabil. 2003 Jan;84(1):29-37. doi: 10.1053/apmr.2003.50061. PMID 12589617
- [Background] Thibaut A, Bodien YG, Laureys S, Giacino JT. Minimally conscious state "plus": diagnostic criteria and relation to functional recovery. J Neurol. 2020 May;267(5):1245-1254. doi: 10.1007/s00415-019-09628-y. Epub 2019 Nov 26. PMID 31773246
- [Background] Wannez S, Heine L, Thonnard M, Gosseries O, Laureys S; Coma Science Group collaborators. The repetition of behavioral assessments in diagnosis of disorders of consciousness. Ann Neurol. 2017 Jun;81(6):883-889. doi: 10.1002/ana.24962. PMID 28543735
- [Background] Kondziella D, Bender A, Diserens K, van Erp W, Estraneo A, Formisano R, Laureys S, Naccache L, Ozturk S, Rohaut B, Sitt JD, Stender J, Tiainen M, Rossetti AO, Gosseries O, Chatelle C; EAN Panel on Coma, Disorders of Consciousness. European Academy of Neurology guideline on the diagnosis of coma and other disorders of consciousness. Eur J Neurol. 2020 May;27(5):741-756. doi: 10.1111/ene.14151. Epub 2020 Feb 23. PMID 32090418